CLINICAL TRIAL: NCT03733236
Title: Implant for Augmentation of Cerebral Blood Flow Trial-1. A Pilot Study Evaluating the Safety and Effectiveness of the Ischemic Stroke System for Treatment of Acute Ischemic Stroke
Brief Title: Safety and Effectiveness Evaluation of the ISS System in Treatment of Acute Ischemic Stroke
Acronym: ImpACT-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BrainsGate (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP1000450
Record Dates: First submitted 2018-11-01; First posted 2018-11-07 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2018-11

CONDITIONS: Ischemic Stricture of Intestine
Keywords: Ischemic Stroke; Treatment; ISS; ImpACT; clinical trial
MeSH Terms: conditions — Ischemic Stroke; Tooth, Impacted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Stimulation (Experimental): The Implant will be implanted using a minimal invasive approach. Following implantation, a CT localization imaging should be performed as soon as possible following the implant procedure. ISS (Ischemic Stroke System) stimulation of the SPG (Sphenopalatine Ganglionduring) for 5 consecutive days.
  Interventions: Device: ISS Active Stimulation

INTERVENTIONS:
Device: ISS Active Stimulation — ISS SPG stimulation and standard of care

SUMMARY:
The primary objective of this pilot study is the assessment of the safety of the ISS500 System in patients who have experienced an acute ischemic stroke within the anterior circulation.

The secondary objectives of this study are to examine the effectiveness of the ISS500 System implantation in the treatment of acute ischemic stroke.

DETAILED DESCRIPTION:
The study is an open label study in which a comparative group of patients will be prospectively selected from a resource of clinical trial data, the Virtual International Stroke Trials Archive (VISTA), on the basis of similar eligibility criteria and match for principal prognostic variables available at trial entry. Data from patients will be transferred to VISTA in a real time or at most, weekly basis and comparative group patients will be prospectively matched throughout the recruitment period. The VISTA investigators will be blinded to treatment group when receiving data from BrainsGate. The VISTA investigators will match each recruited BrainsGate patient with 3 patients from the VISTA archive. The matching criteria will include age ± 4 years; baseline NIH score matched exactly, and side of infarct.

In addition, to the end of treatment visit, in which implanted patients will undergo a device removal procedure, two follow-up visits will be performed. The visits should be performed at 30±5, and at 90±5 post enrollment. Aggregate trial duration will be ~100 days per patient, and the overall study duration will be up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years and ≤ 85 of both genders
2. Patients with symptoms and signs of an acute ischemic hemispheric stroke within the anterior circulation.
3. NIHSS ≥ 7 and ≤ 20
4. Treatment can be initiated within the first 24 hours following stroke onset or since last seen normal.
5. Signed informed consent has been obtained from the patient him/herself or his/her legally authorized representative

Exclusion Criteria:

1. Time interval since onset of symptoms undetermined
2. Treatment with ISS500 System can't start within the first 24 hours post stroke onset
3. Any other imaging diagnosis including tumor, abscess, primary intracranial hemorrhage (ICH) or secondary hemorrhage (PH1-PH2) (H1 and H2 are allowed); or symptoms suspicious for sub-arachnoid hemorrhage, etc
4. Clinical syndrome of an acute stroke due to lacunar infarct (pure motor hemiparesis, ataxic hemiparesis, sensorimotor stroke), unless brain imaging demonstrates a relevant lesion > 1.5 cm in size
5. Not a stroke in the anterior circulation
6. Minor stroke with non-disabling deficit or rapidly improving neurological symptoms with a high probably to Transient Ischemic Attack (TIA)
7. Eligible to or treated with IV or IA t-PA or mechanical thrombolysis
8. Baseline NIHSS >20 or < 7
9. Neurological deficit that has led to stupor or coma (NIHSS level of consciousness score greater than or equal to 2)
10. History of stroke in previous 6 months
11. Pre-existing disability; Modified Rankin Score > 2 upon screening
12. Patients under oral anticoagulants or having received heparin within 48 hours, and / or with elevated activated partial thromboplastin time (aPTT) (or INR)
13. High clinical suspicion of septic embolus
14. Severe cardiac disease: evidence of congestive heart failure or has history of endstage cardiovascular disease (e.g. CHF NYHA Class III or IV or unstable angina)
15. Uncontrolled hypertension upon enrollment (systolic >185 mmHg and/or diastolic >110 mmHg)
16. Serious systemic infection
17. Women known to be pregnant or having a positive or indeterminate pregnancy test
18. Patients with other implanted neural stimulator
19. Orthodontics or non-Hygienic condition/ problems that prevent procedures within the mouth
20. MRI2 contraindications, such as but not limited to:

    * Central nervous system aneurysm clips
    * Implanted cardiac pacemaker or defibrillator;
    * Cochlear implant
    * Ocular foreign body (e.g. metal shavings)
    * Insulin pump
    * Metal shrapnel or bullet
    * Any implanted device that is incompatible with MRI.
    * Patients with a condition precluding entry into the scanner (e.g. morbid obesity, claustrophobia, etc.)
21. Life expectancy < 1 year from other causes
22. Currently participating in any other clinical trial
23. Patients unable or unwilling to follow protocol requirements
24. Massive stroke, defined as acute parenchymal hypodense lesion or effacement of cerebral sulci in over a 2/3 of the MCA territory per CT (or equivalent per T2/Flair/DWI MRI)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-07-06 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Treatment successful completion | 5 Days
  The need to stop the treatment sessions completely or alternately.
Adverse Events profile at 90 Day compared to VISTA trials data | 90 Days
  Adverse Events profile at 90 days post implantation will be compared to the data retrieved form the VISTA trials.

SECONDARY OUTCOMES:
The distribution of modified Rankin scale scores at 90 days | 90 Days
  Shift in the distribution of modified Rankin Scale (mRS) scores at 90 days Favorable outcome is mRS score between 0 and 2
NIHSS scores at 90 days | 90 Days
  The distribution of total NIHSS scores at 90 days - binary NIHSS (defined as the proportion of favorable outcomes assessed using the NIHSS scale, where as favorable outcome was a complete recovery (NIHSS 0 or 1) or an improvement by 9 or more points in the NIHSS score
Proportion of patients achieving a Barthel index at 90 days | 90 Days
  The proportion of patients achieving a Barthel index of 95-100 (versus 0-90) at 90 days

OTHER OUTCOMES:
Patient and treatment compliance to the stimulation | 5 Days
  The ability to maintain treatment in each session for the treatment length, and the compliance for the whole treatment period; i.e. each treatment session should be performed for at least 85% of the prescribed regimen

CONTACTS AND LOCATIONS:
Overall Officials: Subash Kaul, Dr., Principal Investigator — Nizam's Institute of Medical Research Punjagutta, Hyderabad.
Locations (2):
- India (2):
  - Postgraduate Institute of Medical Education and Research, Chandigarh
  - Nizam's Institute of Medical Research Punjagutta, Hyderabad., Hyderabad

REFERENCES:
- [Derived] Khurana D, Kaul S, Schneider D, Csanyi A, Adam I, Ichaporia NR, Griewing B, Csiba L, Valikovics A, Puri V, Diener HC, Schwab S, Hetzel A, Bornstein N; ImpACT-1 Study Group. Implant for Augmentation of Cerebral Blood Flow Trial-1 (ImpACT-1). A single-arm feasibility study evaluating the safety and potential benefit of the Ischemic Stroke System for treatment of acute ischemic stroke. PLoS One. 2019 Jul 3;14(7):e0217472. doi: 10.1371/journal.pone.0217472. eCollection 2019. PMID 31269025